CLINICAL TRIAL: NCT01018771
Title: A Prospective, Randomised Study Comparing the Use of Actifuse (Trademark) Advanced Bone Matrix (ABX) Synthetic Bone Substitute With INFUSE (Trademark) on Fusion in Patients Requiring Posterolateral Instrumented Lumbar Fusion
Brief Title: Actifuse ABX Versus INFUSE in Posterolateral Instrumented Lumbar Fusion
Acronym: APPRAISET2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Apatech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP0803PLF; ACTRN12609000548235 (Other: ANZCTR)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Degenerative Disc Disease
Keywords: actifuse; INFUSE; InductOs; DDD; Degenerative disc disease; PLF; posterolateral lumbar fusion; bone substitute; bone graft; synthetic bone substitute; spinal surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actifuse ABX (Experimental): Actifuse ABX bone substitute
  Interventions: Procedure: Actifuse ABX
- INFUSE, plus Mastergraft granules (Active Comparator)
  Interventions: Procedure: INFUSE, plus Mastergraft granules

INTERVENTIONS:
Procedure: Actifuse ABX — bone graft to be used in posterolateral instrumented lumbar fusion
  Arms: Actifuse ABX
Procedure: INFUSE, plus Mastergraft granules — bone graft to be used in posterolateral instrumented lumbar fusion
  Arms: INFUSE, plus Mastergraft granules

SUMMARY:
This is a prospective randomised study.

Primary objective: Evaluation of success rates of Actifuse ABX and INFUSE in achieving bone fusion.

Secondary objectives: Assess clinical outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Have degenerative disc disease of the lumbar spine as indicated by back pain of discogenic/degenerative origin with or without leg pain and has one or more of the following conditions as documented by Plain X-Rays, CT Scan or MRI Scan:

  * Modic changes.
  * High intensity changes in the annulus.
  * Loss of disc height.
  * Decreased hydration of the disc.
  * Canal stenosis with or without Spondylotic slip.
  * Gross facet joint changes requiring fusion for treatment.
  * Have documented annular pathology by other means. (e.g. with discography).
* Have a preoperative Oswestry Back Disability Score of 30 or more.
* Aged 18 to 75 years and skeletally mature at time of surgery.
* Have not responded to non-operative treatment (e.g. bed rest, physical therapy, medications and/or spinal injections) for a period of six months.
* If of childbearing potential, patient is non-pregnant, non-nursing and agrees not to become pregnant for one year following surgery.
* Is will to and able to comply with the study plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

* Has had previous failed attempts at fusion surgery at the involved level(s).
* Has a diagnosis of spinal infection tumour or trauma.
* Requires surgery at more than two (2) levels.
* Has osteoporosis (excluding osteopenia) as evidenced on plain X-rays, CT Scans (or DEXA scan in cases of doubt).
* Is pregnant.
* Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
* Has received drugs that may interfere with bone metabolism within two weeks prior to the planned surgery date (e.g. steroids or methotrexate) excluding routine perioperative, non-steroidal anti-inflammatory drugs.
* Has a history of autoimmune disease.
* Has a history of exposure to injectable collagen implants.
* Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
* Has received treatment with an investigational therapy (device and/or pharmaceutical) within 30 days prior to surgery or such treatment is planned during the 24 months following surgery.
* Has received any previous exposure to any/all BMPs of either human or animal extraction.
* Has a history of allergy to bovine products or a history of anaphylaxis.
* Has a history of any endocrine or metabolic disorder known to affect osteogenesis (e.g. Paget's disease, renal oseodystrophy, Ehlos-Danlos syndrome or Osteogenesis Imperfecta).
* Has any disease that would preclude accurate clinical evaluation (e.g. neuromuscular disease etc).
* Has a primary diagnosis of a spinal disorder other than degenerative disc disease or other conditions as set out in "Inclusions" above at the involved level(s).
* Has a condition that requires postoperative medications that interfere with fusion, such as steroids or prolonged use of non-steroidal anti-inflammatory drugs, excluding routine perioperative, non-steroidal anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation.
* Has overt or active bacterial infection, local or systemic and/or a potential for bacteremia.
* Has presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
* Has a documented metal allergy or intolerance to titanium alloy or cobalt-chrome-molybdenum alloy.
* Who, in the opinion of the Principal Investigator or Co-Investigators, is intellectually unable to co-operate with the study.
* Has chronic or acute renal and/or hepatic failure or prior history of renal or hepatic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fusion, defined as evidence of bridging trabecular bone present at 1 year | 1 year

SECONDARY OUTCOMES:
Improvement in the following clinical outcomes measurements: Pain/Disability as measured by Oswestry Lower Back Pain Questionnaire; Quality of Life as measured by Short Form Health Survey (SF36)and Neurological Status | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Huub Kruewel, Ph.D, Study Director — Director, Medical Affairs
Locations (1):
- Moloney & Associates, Wollongong, Australia